CLINICAL TRIAL: NCT00162812
Title: Prospective Evaluation of Topoisomerase II Alpha Gene Amplification and Protein Overexpression as Markers Predicting the Efficacy of Epirubicin in the Primary Treatment of Breast Cancer Patients
Brief Title: Topoisomerase II Alpha Gene Amplification and Protein Overexpression Predicting Efficacy of Epirubicin
Acronym: TOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Jules Bordet Institute (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); Centre Paul Strauss (Other); Centre Hospitalier du Luxembourg (Other); Clinique Louis Cathy - Baudour - Belgium (Unknown); HIS - Site Etterbeek - Ixelles - Belgium (Unknown); Clinique Saint Pierre Ottignies (Other); Clinique Ste Elisabeth - Namur - Belgium (Unknown); University Hospital of Crete (Other); Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other)
Responsible Party: Veronique D'Hondt, Jules Bordet Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOP Trial; CE1141
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; early breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epirubicin — 100 mg/m² every three weeks (4 cycles) or every two weeks (6 cycles)

SUMMARY:
prospective evaluation of topoisomerase II alpha gene amplification and protein overexpression as markers predicting the efficacy of epirubicin in the primary treatment of breast cancer patients.

DETAILED DESCRIPTION:
Clinical evaluation of topo II a as a predictive marker: Preliminary results from a clinical study suggest that complete remission after treatment with anthracyclines for advanced breast cancer is observed only in case of topo II a gene amplification (7 complete remissions, all in patients with topo II a gene amplified tumors, no complete remissions in patients with a normal or deleted topo II a gene).

Moreover, our group has analyzed the predictive value of topo II a in a population of node-positive breast cancer patients randomly treated either with anthracyclines or with CMF (Belgian cooperative trial). In a first study, topo II a was evaluated by immunohistochemistry, which allows the detection of topo II a protein expression. The results of this study suggested that patients deriving the highest benefit from anthracyclines were those in which topo II a protein is immunostained in more than 10% of tumor cells. The main findings of this study should be seen as hypothesis-generating because of the limited number of patients evaluated (about fifty in each study arm) and because topo II a protein levels depend on gene amplification as well as on tumor proliferation rate. Therefore, topo II a protein expression does not necessarily reflect topo II a gene status.

The second study run by our group was based on the same series of patients evaluated in the first study, but, this time, both HER-2 and topo II a genes were evaluated by fluorescence in-situ hybridization (FISH), which allows the detection of gene aberrations. The main findings of the second study were quite consistent with the pre-clinical data suggesting that only HER-2 amplified/topo II a amplified tumours show great sensitivity to anthracyclines while the efficacy of these same agents in HER-2 amplified/topo II a non-amplified tumors is comparable to the efficacy of other drugs or regimens like CMF.

Nevertheless, although the results reported in this study bring some additional support to the hypothesis of topo II a as a marker predicting the efficacy of anthracyclines, no definitive conclusions can be drawn because of the fairly limited number of patients evaluated, and the retrospective nature of the analyses.

The present study protocol: Supported by "in-vitro" and preliminary "in-vivo" data, briefly summarized above, this study is designed to test prospectively the value of topo II alpha gene amplification and protein overexpression in predicting the efficacy of anthracyclines. To our knowledge this is the only prospective trial worldwide which is attempting to prospectively clarify the predictive value of this interesting biological marker. This study could have important practical implications in the daily clinical management of early breast cancer patients because, if the trial confirms that topo II a gene amplification and/or protein overexpression are associated with high efficacy of anthracyclines, while topo II a normal/deleted gene and low protein content are associated with modest efficacy, an important step forward in the direction of anthracycline "tailoring" would be accomplished.

The practical advantage of this approach would be to use anthracyclines primarily in patients who are supposed to derive the largest benefit, thus sparing the long-term anthracycline-related toxicity (i.e. secondary acute myeloid leukemia, cardiac dysfunction, and amenorrhea/sterility in case of fertile women) to those patients for whom no significant gain in antitumor activity is anticipated.

To reach this ambitious aim, early breast cancer patients with tumors of at least 2 cm (defined by breast ultrasound) will be evaluated for topo II a gene and protein expression. For this purpose, a pre-treatment biopsy (tru-cut) will be performed and topo II a gene will be evaluated on fixed samples by FISH. The use of a triple probe will allow the concomitant evaluation of the HER-2 gene status. Topo II a protein will be evaluated by immunohistochemistry (IHC). Afterwards, all patients, independently of the topo II a gene and protein status, will be treated with single-agent epirubicin Eligibility criteria will allow the participation of patients for whom the use of an anthracycline-based adjuvant therapy would have been most probably proposed after breast cancer surgery, mainly because of estrogen receptor (ER) negativity. Therefore, no overtreatment with anthracyclines will occur in this group of patients. Pathological complete response (pCR) to epirubicin will be correlated with the topo II a gene and protein status. The study has two biological hypotheses, one for the subgroup of patients with ER negative/HER-2 amplified tumors, the other one for the subgroup of patients with ER negative/HER-2 non amplified tumors.

1. st hypothesis: Patients with ER negative/HER-2 amplified tumors: In this subgroup of patients, topo II a gene will be amplified in about 40% of cases. We hypothesize that in topo II a amplified tumors a three-fold increase in pCR rate will be observed, as opposed to the pCR rate in tumors with topo II a normal or deleted gene.
2. nd hypothesis : Patients with ER negative/HER-2 non amplified tumors: In this subset of patients, almost no topo II a gene aberrations will be found based on previous data discussed above. However, recent data reported by C. Sotiriou et al using cDNA microarrays, suggest that in this subset of ER-negative HER-2 negative tumors, also defined as the basal-like subset, two distinct subgroups can be identified (i.e. basal-like 1 and 2). While basal-like 1 tumors show a high proliferation rate and high levels of topo II a RNA, basal-like 2 tumors have a moderate-low proliferation rate and normal levels of topo II a RNA. We hypothesize that the topo II a RNA overexpression in basal-like 1 tumors is not related to topo II a gene amplification because no concomitant HER-2 gene amplification is reported in this subset of tumors. The second study hypothesis is that in ER negative/HER-2 non amplified tumors with topo II a protein overexpression, a 2.5 fold increase in pCR rate will be observed, as opposed to the pCR rate in tumors with low topo II a protein content.

A tumor sample drawn at the time of pre-treatment biopsy will be frozen and used to perform oligonucleotide based microarrays (Affymetrix). This technique allows the evaluation of thousands of genes and ultimately provides us with the tumor genetic profile. Homogeneous genetic profiles (genetic clusters) that might be identified, will be correlated with the efficacy of single-agent epirubicin. This correlation will allow us to address the secondary end-point of this study, which is the identification of other genes or eventually a genetic profile playing a role in the determination of sensitivity to anthracyclines. Among the genes that could interfere with sensitivity to anthracyclines, p-53 seems to deserve special attention. Indeed, "in-vitro" data suggest that at least some p-53 mutated tumors are poorly sensitive to anthracyclines, primarily because anthracycline-induced apoptosis is prevented. Interestingly, p-53 mutated tumors display frequently HER-2 gene amplification and therefore topo II a gene amplification (23). Accordingly, p-53 mutations could hamper response to anthracyclines even in tumors carrying topo II a gene amplification. This hypothesis will also be explored in the present study, because p-53 mutations will be evaluated by DNA sequencing, and the efficacy of epirubicin in topo II a amplified and non-amplified tumors will be correlated with p-53 status.

Additionally, patients with inflammatory breast cancer will be treated with dense administration of epirubicin (100 mg/m2/2 weeks). We keep the same drug as for early breast cancer but we use a slightly more aggressive regimen with a higher dose-density. The feasibility of the administration of epirubicin 100 mg/m2 every two weeks with granulocyte-growth factor support has been shown in the neoadjuvant, metastatic and adjuvant settings with acceptable toxicity. This neoadjuvant epirubicin regimen may be completed by adjuvant chemotherapy, such as taxane-based regimens, since the sequential approach (anthracyclines and taxanes) has been suggested superior to anthracyclines regimen in LABC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed breast cancer (operable, locally advanced or inflammatory)
2. Age less than 70 years
3. Female patient
4. Tumor size 2 cm at ultrasound examination.
5. ER-negative tumors defined according to immunohistochemistry (i.e. < 10% of positive cells after immunostaining).
6. Multifocal and multicentric breast tumors are allowed if all foci are ER-negative.
7. Fixed and frozen samples from the primary tumor, obtained before treatment with epirubicin, must be available for evaluation of biological markers (topo II alpha gene and protein, HER-2 gene, p-53 gene, oligonucleotides microarrays).
8. Written informed consent before study registration.
9. Performance status 0 or 1 (ECOG scale)
10. Normal CBC, hepatic and renal functions
11. Normal left ventricular ejection fraction by echocardiography or muga scan
12. Negative pregnancy test for all women of childbearing potential. Patients of childbearing potential must implement adequate non-hormonal measures to avoid pregnancy during treatment.

Exclusion Criteria:

1. Metastatic breast cancer
2. Serious medical conditions like:

   1. congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled arrhythmias.
   2. history of significant neurologic or psychiatric disorders
   3. active uncontrolled infection
   4. active peptic ulcer, unstable diabetes mellitus
3. Concomitant contralateral invasive breast cancer
4. Concurrent treatment with hormonal replacement therapy
5. Concurrent treatment with any other anti-cancer therapy
6. Previous treatment with anthracyclines for breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2003-01; Primary Completion 2008-12 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
correlation of topoisomerase II and pathologic complete response | pCR at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Veronique D'Hondt, MD, PhD, Principal Investigator — Jules Bordet Institute; Martine Piccart, MD, PhD, Study Chair — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium